CLINICAL TRIAL: NCT00030485
Title: A Phase II Study of OSI-774 (NSC 718781) in Patients With Locally Advanced and/or Metastatic Carcinoma of the Endometrium
Brief Title: Erlotinib in Treating Patients With Locally Advanced and/or Metastatic Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NCIC Clinical Trials Group (Network)
Purpose: Treatment
Other Study IDs: I148; CAN-NCIC-IND148; NCI-NCIC-148; CDR0000069169 (Other: PDQ)
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Endometrial Cancer
Keywords: stage IV endometrial carcinoma; recurrent endometrial carcinoma; endometrial adenocarcinoma; endometrial adenosquamous cell carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Erlotinib Hydrochloride

INTERVENTIONS:
Drug: erlotinib hydrochloride

SUMMARY:
RATIONALE: Biological therapies such as erlotinib may interfere with the growth of tumor cells and slow the growth of the tumor.

PURPOSE: Phase II trial to determine the effectiveness of erlotinib in treating patients who have locally advanced and/or metastatic endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of erlotinib, in terms of response rate and duration of stable disease, in patients with locally advanced and/or metastatic carcinoma of the endometrium.
* Determine the toxicity of this drug in these patients.
* Determine the time to progression and duration of response in patients treated with this drug.
* Correlate objective tumor response with levels of epidermal growth factor receptor expression in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral erlotinib once daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 weeks. Patients with complete or partial response or stable disease are also followed every 3 months until relapse or death.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic and/or locally advanced adenocarcinoma or adenosquamous carcinoma of the endometrium

  * Incurable by standard therapies
* Clinically and/or radiologically documented disease with at least 1 unidimensionally measurable site

  * At least 20 mm by x-ray, physical exam, or CT scan OR
  * At least 10 mm by spiral CT scan
  * Bone metastases considered nonmeasurable
* Tumor tissue from primary tumor available for assessing epidermal growth factor receptor (EGFR) status
* No uterine sarcomas (leiomyosarcoma), mixed mullerian tumors, and/or adenosarcomas
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Platelet count at least 100,000/mm3
* Absolute granulocyte count at least 1,500/mm3

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina
* No cardiac arrhythmia

Gastrointestinal:

* No gastrointestinal (GI) tract disease that would preclude ability to take oral medication
* No requirement for IV alimentation
* No uncontrolled inflammatory GI disease (e.g., Crohn's disease or ulcerative colitis)
* No active peptic ulcer disease

Ophthalmic:

* No significant ophthalmologic abnormalities, including any of the following:

  * Prior severe dry eye syndrome, Sjogren's syndrome, or keratoconjunctivitis sicca
  * Severe-exposure keratopathy
  * Disorders that would increase the risk of epithelium-related complications (e.g., bullous keratopathy, aniridia, severe chemical burns, or neutrophilic keratitis)
  * Congenital abnormality (e.g., Fuch's dystrophy)
  * Abnormal slit-lamp examination using a vital dye (e.g., fluorescein or Bengal-Rose)
  * Abnormal corneal sensitivity test (e.g., Schirmer test or similar tear production test)
* No concurrent ocular inflammation or infection

Other:

* No other malignancy within the past 5 years except adequately treated nonmelanoma skin cancer or curatively treated carcinoma in situ of the cervix
* No prior allergic reaction attributed to compounds of similar biological or chemical composition to erlotinib
* No other concurrent serious illness or medical condition that would preclude study
* No prior significant neurologic or psychiatric disorder that would preclude study
* No active uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for endometrial cancer

Endocrine therapy:

* No more than 1 prior hormonal therapy (progestational agent or aromatase inhibitor) in the adjuvant or metastatic setting
* At least 1 week since prior hormonal therapy

Radiotherapy:

* At least 4 weeks since prior radiotherapy (except for low-dose palliative radiotherapy) and recovered

Surgery:

* At least 3 weeks since prior major surgery and recovered
* No prior surgical procedures affecting absorption
* No concurrent ophthalmic surgery

Other:

* No prior EGFR-targeting therapies
* No other concurrent investigational therapy
* No other concurrent anticancer therapy
* Concurrent oral anticoagulants (e.g., warfarin) allowed provided there is increased vigilance with respect to monitoring INR
* Concurrent low molecular weight heparin allowed at investigator's discretion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit M. Oza, MD, Study Chair — Princess Margaret Hospital, Canada
Locations (8):
- Canada (8):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Notre- Dame du CHUM, Montreal, Quebec

REFERENCES:
- [Result] Oza AM, Eisenhauer EA, Elit L, Cutz JC, Sakurada A, Tsao MS, Hoskins PJ, Biagi J, Ghatage P, Mazurka J, Provencher D, Dore N, Dancey J, Fyles A. Phase II study of erlotinib in recurrent or metastatic endometrial cancer: NCIC IND-148. J Clin Oncol. 2008 Sep 10;26(26):4319-25. doi: 10.1200/JCO.2007.15.8808. Epub 2008 Jun 30. PMID 18591547
- [Result] Oza A, Elit L, Eisenhauer E, et al.: Phase II study of erlotinib (Tarceva, OSI 774) in women with recurrent or metastatic endometrial cancer -- NCIC IND.148. [Abstract] Clin Cancer Res 9 (Suppl): A-105, 6094s, 2003.